CLINICAL TRIAL: NCT03406676
Title: The Preventive Effects of Pre-treatment With Methylene Blue for Vascular Paralysis of the Patients With Obstructive Jaundice During Operation
Brief Title: Pre-treatment With Methylene Blue Prevent Peri-operative Reduced Systemic Vascular Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shuguo Zheng, MD, Professor of Institute of Hepatobiliary Surgery, Southwest Hospital, Third Military Medical University Affiliation: Southwest Hospital, China, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MZK002
Record Dates: First submitted 2018-01-04; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Obstructive Jaundice
Keywords: Methylene blue; Peripheral vascular resistance
MeSH Terms: conditions — Jaundice, Obstructive | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene blue (Experimental): 2mg / Kg of methylene blue in volume of 50ml is administrated I.V before anesthesia induction.
  Interventions: Drug: Methylene Blue
- saline (No Intervention): 50ml of saline is administrated I.V before anesthesia induction.

INTERVENTIONS:
Drug: Methylene Blue — 2mg / Kg of methylene blue in volume of 50ml is administrated I.V before anesthesia induction.
  Other Names: Methylene blue injection
  Arms: Methylene blue

SUMMARY:
To explore the effects of pre-treatment with methylene blue on reduced perioperative vascular resistance in patients with obstructive jaundice.

DETAILED DESCRIPTION:
Hemodynamic characteristics of patients with obstructive jaundice are high cardiac output, low peripheral vascular resistance. The molecular basis for this feature is the increased production of NO. Methylene blue can increase peripheral resistance, the mechanism is: methylene blue is an oxidoreductase inhibitor, can inhibit the increased production of NO in the vascular endothelium, thereby increasing peripheral vascular resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18-60 years;
2. American Society of Anesthesiologists（ASA） grade I~III;
3. TBIL>ULN and TBA>ULN; The patients with obstructive jaundice.

Exclusion Criteria:

1. Organs dysfunction(heart,lungs and etc);
2. Mental disorders;
3. in other clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Peripheral vascular resistance | through operation completion, an average of 6 hours
  the dose of vasoconstrictors used to Maintain Peripheral vascular resistance in the normal range (800 ~ 1200dyns / cm5)

CONTACTS AND LOCATIONS:
Overall Officials: Zheng ShuGuo, Principal Investigator — MD Study Director Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China